CLINICAL TRIAL: NCT06620952
Title: Effect of the "O-ring" Technique in Reducing Cerebrospinal Fluid Leak in Posterior Fossa Surgery: an Explorative Study
Acronym: O'Ring
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Francesco Guerrini, Doctor, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: O'Ring
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Posterior Fossa Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients operated for a disease located in posterior fossa: Patients operated for a disease located in posterior fossa for which a RS, KR or CH approach has to be performed. Patients between January 2018 and October 2023 will be considered for the study. Lacking of clinical, radiological and surgical data represe
  Interventions: Procedure: O-ring technique

INTERVENTIONS:
Procedure: O-ring technique — "O-ring technique." consists on a different arrangement of fibrin-glue on a polymethilmetacrylate cranioplasty, with the aim to create a gasket to prevent CSF leakage

SUMMARY:
Posterior fossa surgery represents on of the most demanding procedure in neurosurgery. Retrosygmoid (RS), key-hole retrosygmoid (KR) and cerebellar hemispheric (CH) are the most common approaches used to access in this area. Despite they are not technically difficult to perform, these approaches can be burdened by postoperative cerebrospinal fluid (CSF) leakage, both at short and long-term follow-up, with an high risk of meningitis. Many techniques were employed to avoid this risk, but it can still be estimated between 2% and 11% according to literature1-4. Spena et al. reported a CSF leakage rate of 6.8% in a previous experience5. As a consequence, newer efforts are necessaries to avoid this potentially lethal complication. By this explorative study, we want to retrospectively analyzed our experience with a newer technique of bone closure, called O'Ring, in patients subdued to posterior fossa surgery by RS, KR and CH approaches, focusing on postoperative CSF leakage (primary objective), wound complications and subcutaneous CSF collections (secondary objectives).

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years,
* availability of pre- and postoperative radiological and clinical data,
* a follow-up period of at least 3 months.

Exclusion Criteria:

* Lacking of clinical, radiological and surgical data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated for a disease located in posterior fossa for which a RS, KR or CH approach has to be performed. Patients between January 2018 and October 2023 will be considered for the study.Lacking of clinical, radiological and surgical data represented exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2024-07-16 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
to estimate incidence of postoperative CSF leakage | 7 days
  cumulative incidence of postoperative CSF leakage

SECONDARY OUTCOMES:
to estimate incidence CSF leakage at 1- and 3-months of follow-up. | 1 and 3 months
  cumulative incidence of CSF leakage at 1- and 3-months follow-up
to estimate the incidence of wound complications postoperatively and at 1- and 3-months | 1 and 3 months
  cumulative incidence of wound complications postoperatively and at 1- and 3-months follow-up
to estimate the incidence of subcutaneous CSF collections postoperatively and at 1 and 3-months radiological follow-up | 1 and 3 months
  cumulative incidence of subcutaneous CSF collections postoperatively and at 1 and 3-months radiological follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- SC Neurochirurgia, Fondazione IRCCS Policlinico San Matteo, Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No